CLINICAL TRIAL: NCT06108518
Title: Clinical Study Evaluating the Effect of Carvedilol in Patients With Active Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Yomna Abdelrafea Ahmed, Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Carvedilol in active RA
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Carvedilol; Hypertension
MeSH Terms: conditions — Arthritis, Rheumatoid; Hypertension | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: randomized, double blind placebo controlled parallel study
Who Masked: Participant, Investigator
Masking Description: The blindness will be maintained by the similarity between the placebo and carvedilol tablets. The patients will be randomized by a neutral researcher using sealed envelope method with assigned code into two groups
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): Group1 (Placebo group; n=35) which will receive the standard treatment for RA plus placebo tablet for 3 months.
  Interventions: Drug: Carvedilol
- Treatment group (Active Comparator): Group 2 (Carvedilol group; n=35) which will receive the standard treatment for RA plus carvedilol 12.5mg once a day for 2 days; this is increased to 25 mg once a day or 12.5 mg twice a day for 3 months.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Treatment group will take carvedilol 12.5mg once a day for 2 days; this is increased to 25 mg once a day or 12.5 mg twice a day for 3 months.

SUMMARY:
This study aims at investigating the possible efficacy and safety of carvedilol as an adjunctive therapy in patients with active rheumatoid arthritis and hypertension.

DETAILED DESCRIPTION:
heumatoid arthritis (RA) is a chronic systemic autoimmune disease that primarily affects the lining of the synovial joints and is associated with progressive disability, premature death, and socioeconomic burdens. It is characterized with chronic production of pro-inflammatory cytokines, which lead to cartilage and bone degradation that results in tissue destruction by the patients' immune system (Guo et al., 2018).

The high systemic inflammatory burden associated with RA appears to be a key driver of increased CV risk. This inflammatory state is linked to endothelial dysfunction and accelerated atherosclerosis (Giollo et al., 2018). Consequently, RA increases the risk of cardiovascular (CV) mortality by up to 50% compared with the general population and CV disease is the leading cause of death in RA patients. This leads to suggestion that reducing inflammation lowers CV risk in RA (Dijkshoorn et al., 2022).

Therapies targeting inflammation remain the mainstay of RA treatment such as non- steroidal anti-inflammatory drugs (NSAIDs), non-biologic and biologic disease-modifying anti-rheumatic drugs (DMARDs), immune-osuppressants, and corticosteroids. However, current treatment strategies have many adverse effects and a significant proportion of RA patients did not effectively respond to them (Aletaha and Smolen., 2018). Consequently, it is crucial to find new therapeutic approaches for the management of inflammation as well as the prevention of cardiovascular complications in rheumatoid arthritis patients.

Carvedilol is a non-selective β-blocker with α-adrenergic receptor antagonism properties which has been safely used in treatment of several cardiovascular disorders (Prajapati et al., 2017). Previous animal studies highlights evidences for the promising anti- arthritic effects of carvedilol that could be mediated through attenuation of leukocyte migration, alleviation of oxidative stress and suppression of pro-inflammatory cytokines such as tumor necrosis factor-α (TNF-α) and interlukin-6 (IL-6) and eicosanoids including prostaglandin E2 (PGE2) and leukotriene B4 (LTB4) (Arab and El-Sawalhi, 2013; Ahmed et al., 2017; Osman et al., 2017).

Taken together, carvedilol has powerful antioxidant/anti-inflammatory properties; we aimed to investigate its protective potential against arthritis that may add further benefits for its clinical usefulness especially in RA patients with concomitant cardiovascular disorders

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis (not in remission) according to American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 criteria i.e 28 joints disease activity score (DAS-28) >2.6.
* Patients with hypertension who are candidate to carvidolol.
* Age range between 18 and 60 years old.
* The studywillbecarriedoutbetween June 2023 and June 2025.
* Both sexes.
* Sex ratio, body mass index (BMI), age, disease activity, and disease duration matched patients.
* Patients receive matched doses of standard treatment including methotrexate, non-steroidal anti-inflammatory drugs, selective cyclooxygenase-2 inhibitors, acetaminophen, and low dose of oral corticosteroids (prednisolone < 15 mg) will be allowed to be enrolled the trial.
* Intravenous, intra-articular or intramuscular corticosteroids; intra-articular hyaluronate sodium and biological DMARDs will not be permitted less than 4 weeks before the first dose of carvedilol.

Exclusion Criteria:

* Patients with congestive heart failure, other heart disease (arrhythmia, ischemic heart disease including angina and myocardial infarction).
* Patients with other inflammatory diseases and active infection.
* Patients with glaucoma.
* Patients with asthma, COPD, other lung diseases.
* Patients with hepatic and biliary diseases.
* Patients with chronic renal failure or those on dialysis.
* Patients with peripheral intermittent claudication and peripheral circulatory disorders.
* Patients receiving oral pednisolone greater than 15 mg/day.
* Patients receiving biological DMARDs.
* Patients with hypersensitivity to carvedilol.
* Patients using antioxidants.
* Pregnant and lactating females.
* Patients receiving digitalis, anti-arrhythmic (amiodarone, propafenone) MAOI, cyclosporine, calcium channel blockers (verapamil, deltiazem), beta blockers, other antihypertensive medications hepatic microsomal enzymes inducers or inhibitors (phenytoin, rifampin, valoproate), oral hypoglycemic and insulin to avoid potential pharmacodynamics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
change in DAS-28-CRP score and the Multidimensional Health Assessment Questionnaire (MDHAQ) scores. | 12 week
  By the end of the study we should notice decrease in DAS-28-CRP score and the Multidimensional Health Assessment Questionnaire (MDHAQ) scores.

SECONDARY OUTCOMES:
change in the serum level of the assessed biological markers | 12 week
  By the end of the study we should notice decrease in serum level of the assessed biological markers
  * C-reactive protein (CRP).
  * 8-hydroxydeoxyguanosine (8-OHdG).
  * Interlukin-6 (IL-6).
  * Leukotriene B4 (LTB4

CONTACTS AND LOCATIONS:
Overall Officials: Dr/Tarek Mohamed, Professor, Study Director — Tanta University

REFERENCES:
- [Background] Ahmed YM, Messiha BA and Abo-Saif AA. Granisetron and carvedilol can protect experimental rats against adjuvant-induced arthritis. Immunopharmacol Immunotoxicol., 2017; 39(2):97-104. Aletaha D, and Smolen JS. Diagnosis and Management of Rheumatoid Arthritis: A Review. JAMA. 2018; 320 (13):1360-1372. Aletaha D, Neogi T, Silman AJ, et al. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010;62(9):2569-2581. Arab HH and El-Sawalhi MM. Carvedilol alleviates adjuvant-induced arthritis and subcutaneous air pouch edema: Modulation of oxidative stress and inflammatory mediators. Toxicol Appl Pharmacol., 2013;268(2):241-248. Dijkshoorn B, Raadsen R and Nurmohamed MT. Cardiovascular Disease Risk in Rheumatoid Arthritis Anno 2022. J Clin Med., 2022 ;11(10):2704. El Miedany Y, El Gaafary M, Youssef SS, et al. Validity of the Developed Arabic Multidimensional Health Assessment Questionnaire for use in standard clinical care of patients with rheumatic diseases. Int J Rheum Dis., 2008; 11:224-236. Giollo A, Bissell LA and Buch MH. Cardiovascular outcomes of patients with rheumatoid arthritis prescribed disease modifying anti-rheumatic drugs: A review. Expert Opin Drug Saf., 2018 ;17(7):697-708. Guo Q, Wang Y, Xu D, et al. Rheumatoid arthritis: Pathological mechanisms and modern pharmacologic therapies. Bone Res., 2018; 6:15.